CLINICAL TRIAL: NCT06830759
Title: EpcoReal: A Multi-country, Prospective Observational Study of Epcoritamab in NHL Comprising Two Patient Cohorts (3L+ (D)LBCL and 3L+ FL)
Brief Title: Real-World Study to Assess Subcutaneous Epcoritamab in Adult Participants With Diffuse Large B-Cell and Follicular Lymphoma
Acronym: EpcoReal
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-903
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-cell Lymphoma; Follicular Lymphoma
Keywords: Diffuse large B-cell lymphoma; Follicular Lymphoma; Epcoritamab
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Epcoritamab: Participants will receive epcoritamab as prescribed by their physician according to local label.

SUMMARY:
Diffuse large B-cell lymphoma (DLBCL) is an aggressive and rare cancer of a type of immune cells (a white blood cell responsible for fighting infections) and the most common type of non-Hodgkin lymphoma. Follicular Lymphoma (FL) is a slow-growing type of non-Hodgkin lymphoma. The purpose of this study is to assess the real-world effectiveness of subcutaneous epcoritamab in adult participants with advanced DLBCL and FL.

Epcoritamab is an investigational drug being developed for treating participants with DLBCL and FL. Approximately 700 participants will be enrolled in approximately 80 sites across 12-20 countries globally.

Participants will receive epcoritamab as prescribed by their physician in accordance with local country label. Participants will be followed for up to 3 years.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are scheduled to be treated with epcoritamab for Treatment after two or more prior lines of therapy 3L+ diffuse large B-cell lymphoma ((D)LBCL) or 3L+ Follicular lymphoma (FL).
* Treatment with epcoritamab should be administered in accordance with the approved local label in the participating country.
* The decision to treat the participant should have been made by the clinician prior to, and independently of any decision to approach the participant to participate in this study.

Exclusion Criteria:

* Any condition included in the contraindications section of the approved local epcoritamab label in the participating country.
* Participation in a concurrent interventional clinical trial (not including non-interventional/ observational study, PMOS, or registry participation) from enrollment and throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants who are being treated with epcoritamab for Diffuse Large B-Cell and Follicular Lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2031-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Overall Response (OR) | Up to approximately 3 years
  Defined as the percentage of participants who achieve best overall response of complete response (CR) or partial response (PR) determined by Lugano criteria

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (63):
- Argentina (6):
  - Hospital Britanico de Buenos Aires /ID# 274419, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Hospital Universitario Austral /ID# 274393, Pilar, Buenos Aires
  - Instituto Alexander Fleming /ID# 277284, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Hospital Privado Universitario De Córdoba /ID# 274457, Córdoba, Córdoba Province
  - Hospital Italiano de Buenos Aires /ID# 274418, Buenos Aires
  - Fundacion Argentina contra la Leucemia (FUNDALEU) /ID# 274390, Buenos Aires
- Austria (2):
  - Krankenhaus Der Barmherzigen Brueder Graz /ID# 273288, Graz, Styria
  - Landeskrankenhaus Hochsteiermark, Standort Leoben /ID# 273266, Leoben, Styria
- Belgium (9):
  - Algemeen Ziekenhuis klina /ID# 273405, Brasschaat, Antwerpen
  - Universitair Ziekenhuis Brussel /ID# 273403, Jette, Brussels Capital
  - Centre Hospitalier Epicura - Hornu /ID# 273406, Boussu, Hainaut
  - Grand Hôpital De Charleroi - Notre Dame /ID# 273728, Charleroi, Hainaut
  - Helora /ID# 273726, La Louvière, Hainaut
  - Groupe Sante CHC - Clinique du MontLegia /ID# 273407, Liège, Liege
  - Ziekenhuis Oost-Limburg, Campus St.-Jan /ID# 273729, Genk, Limburg
  - Vitaz /Id# 273408, Sint-Niklaas, Oost-Vlaanderen
  - AZ Oostende /ID# 273714, Ostend, West-Vlaanderen
- Bulgaria (4):
  - Umhat Sveti Ivan Rilsky /ID# 274898, Sofiya, Sofia
  - University Multiprofile Hospital for Active Treatment Dr. Georgi Stranski /ID# 274893, Pleven
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 273659, Sofia
  - Specialized Hospital For Active Treatment Of Haematology Diseases /ID# 274955, Sofia
- Canada (5):
  - Cross Cancer Institute /ID# 271504, Edmonton, Alberta
  - The Moncton Hospital /ID# 277230, Moncton, New Brunswick
  - Eastern Health - General Hospital /ID# 272062, St. John's, Newfoundland and Labrador
  - Health Sciences North /ID# 274738, Greater Sudbury, Ontario
  - Kingston General Hospital /ID# 272061, Kingston, Ontario
- Greece (11):
  - Agios Andreas Hospital Patras /ID# 273629, Pátrai, Achaia
  - Evangelismos Hospital /ID# 272736, Athens, Attica
  - General Hospital of Athens Laiko /ID# 272758, Athens, Attica
  - University General Hospital Attikon /ID# 272738, Athens, Attica
  - Metaxa Cancer Hospital Of Piraeus /ID# 273623, Piraeus, Attica
  - University General Hospital of Alexandroupoli /ID# 272737, Alexandroupoli, Evros
  - University Hospital of Ioannina /ID# 272739, Ioannina
  - AHEPA University General Hospital of Thessaloniki /ID# 273633, Thessaloniki
  - General Hospital of Thessaloniki Hippokrateio /ID# 273635, Thessaloniki
  - Papageorgiou General Hospital /ID# 272735, Thessaloniki
  - General Hospital Of Thessaloniki G. Papanikolaou /ID# 275323, Thessaloniki
- Israel (3):
  - Tel Aviv Sourasky Medical Center /ID# 271615, Tel Aviv, Tel Aviv
  - Hadassah Medical Center-Hebrew University /ID# 271616, Jerusalem
  - Rabin Medical Center. /ID# 271614, Petah Tikva
- Italy (4):
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli /ID# 274215, Naples, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 274572, Rome, Roma
  - I.R.C.C.S Istituto Tumori Giovanni Paolo II /ID# 274217, Bari
  - Ospedale La Maddalena /ID# 274411, Palermo
- Hematologica Alta Especialidad /ID# 275279, Huixquilucan de Degollado, Mexico
- Portugal (2):
  - Unidade Local de Saude de Coimbra, EPE /ID# 272720, Coimbra
  - Unidade Local de Saúde Trás-os-Montes e Alto Douro /ID# 275404, Vila Real
- Spain (12):
  - Complejo Hospitalario Universitario A Coruña /ID# 272040, A Coruña, A Coruna
  - Institut Català d'Oncologia (ICO) - Badalona /ID# 272043, Badalona, Barcelona
  - Hospital Universitari Parc Tauli /ID# 272044, Sabadell, Barcelona
  - Hospital Universitario Reina Sofia /ID# 272051, Córdoba, Cordoba
  - Hospital Costa del Sol /ID# 272431, Marbella, Malaga
  - Hospital Universitario de Navarra /ID# 272041, Pamplona, Navarre
  - Hospital Universitario de Valme /ID# 272050, Seville, Sevilla
  - Hospital de Manises /ID# 272046, Manises, Valencia
  - Hospital Universitario De Burgos /ID# 272066, Burgos
  - Hospital General Universitario Morales Meseguer /ID# 272466, Murcia
  - Hospital Universitario Nuestra Señora de Candelaria /ID# 272413, Santa Cruz de Tenerife
  - Hospital Clinico Universitario de Valladolid /ID# 272042, Valladolid
- United Kingdom (4):
  - Milton Keynes Hospital /ID# 272817, Milton Keynes, Buckinghamshire
  - Royal Cornwall Hospital /ID# 272747, Truro, Cornwall
  - Cheltenham General Hospital /ID# 272746, Cheltenham, Gloucestershire
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 272748, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-903